CLINICAL TRIAL: NCT07151599
Title: Randomized Controlled Trial Comparing Fractional Erbium:Glass (1540-1550 nm) and Thulium (1927 nm) Lasers Versus Microneedling for the Treatment of Atrophic Acne Scars
Brief Title: Efficacy of Combined Fractional Er:Glass and Thulium Lasers Versus Microneedling for Atrophic Acne Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Christiane Pavani, Randomized Controlled Trial Comparing Combined Fractional Erbium:Glass and Thulium Lasers Versus Microneedling for the Treatment of Atrophic Acne Scars, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ErGlass_MedicinaBiofotonica
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acne Scars
Keywords: Fractionated Erbium Glass Laser; Fractionated Thulium Laser; Microneedling; Percutaneous Induction of Collagen; Acne Scars
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Participants are assigned to Microneedling or Combination of Thulium and Erbium Glass Fractionated Laser in parallel.
Who Masked: Outcomes Assessor
Masking Description: Assesor evaluation of the outcomes will be performed in anonymous pictures. The participant reported outcomes will not be blinded, since participant will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedling (Active Comparator): Microneedling performed with an electronic pen and sterile disposable cartridge of 12 needles at 2mm depth
  Interventions: Device: Microneedling
- Fractionated Er:Glass and Thulium Lasers (Experimental): Fractional Erbium:Glass laser is applied first, focused on scarred areas, followed immediately by fractional Thulium 1927 nm over the full face.
  Interventions: Device: Fractionated Er:Glass Laser combined to Fractionated Thulium Laser

INTERVENTIONS:
Device: Microneedling — Microneedling performed with an electronic pen and sterile disposable cartridge with 12 needles and 2mm depth, three treatment sessions at four-week intervals.
  Arms: Microneedling
Device: Fractionated Er:Glass Laser combined to Fractionated Thulium Laser — Fractional Erbium:Glass laser will be applied first, focused on scarred areas (50 mJ, 15 ms e 100 PPA) , followed immediately by fractional Thulium 1927 nm over the full face (10 mJ, 1 ms e 100 PPA), three treatment sessions at four-week intervals.
  Arms: Fractionated Er:Glass and Thulium Lasers

SUMMARY:
The purpose of this study is to compare two treatments for acne scars on the face. The study will test whether fractional lasers (Erbium:Glass and Thulium) lead to better improvement in acne scars than microneedling.

DETAILED DESCRIPTION:
Acne scars are common and can have a lasting impact on self-esteem, social relationships, and quality of life. Several treatment options exist, but many patients continue to seek better results. Microneedling is a minimally invasive technique that uses small needles to stimulate skin repair. Fractional lasers, such as Erbium:Glass (1540-1550 nm) and Thulium (1927 nm), deliver energy into the skin to promote remodeling of deeper and more superficial layers. The combination of these two fractional lasers may provide a more comprehensive treatment approach for acne scars.

This clinical trial will directly compare these two options: microneedling versus the combined use of fractional Erbium:Glass and Thulium lasers. A total of 84 adults between 18 and 30 years old with atrophic acne scars will take part. Participants will be randomly chosen by a draw (like a lottery) to receive one of the two groups. Both groups will receive three treatment sessions, with four weeks between each session.

The main goal is to determine which treatment leads to greater improvement in acne scars. Improvement will be measured by independent evaluators who will compare standardized before-and-after photographs using a grading scale. Participants will also report their own satisfaction with the results and how well they tolerated the treatments. Follow-up assessments will occur up to 90 days after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin phototypes I to VI
* Presence of atrophic acne scars on the face

Exclusion Criteria:

* Decompensated systemic diseases
* Any active infection (e.g., viral such as herpes, bacterial, or fungal)
* Pregnant or breastfeeding women
* Presence of hypertrophic or keloid scars
* Current use of anticoagulant or antiplatelet medications
* History of hemophilia or coagulation disorders
* Current use of anti-inflammatory drugs or corticosteroids
* Use of retinoids, including isotretinoin, within the past 6 months
* Exposure to sunlight within the past 15 days
* Undergoing any aesthetic facial treatment or having undergone scar treatments in the facial region within 180 days prior to study initiation
* Presence of active acne (occasional isolated lesions will not be considered exclusion criteria)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — cisgender women and cisgender men
Enrollment: 84 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
ECCA grading scale (échelle d'évaluation clinique des cicatrices d'acné) | Assessments will be performed by blinded evaluators using standardized photographs at baseline.
  The ECCA is a validated scale that quantifies acne scars through both qualitative and quantitative components. Scar type is weighted by a numerical factor (15-30 for atrophic scars and elastosis; 40-50 for hypertrophic/keloid scars) and multiplied by the number of lesions, graded on a 4-point scale: 0 = none; 1 = <5 scars; 2 = 5-20 scars; 3 = >20 scars. The global score ranges from 0 to 540, with higher scores indicating greater severity. In this study, participants with hypertrophic or keloid scars will be excluded; therefore, only atrophic scar subtypes will be scored (subcategory 1).
ECCA grading scale (échelle d'évaluation clinique des cicatrices d'acné) | Assessments will be performed by blinded evaluators using standardized photographs at 30 days after the last session.
  The ECCA is a validated scale that quantifies acne scars through both qualitative and quantitative components. Scar type is weighted by a numerical factor (15-30 for atrophic scars and elastosis; 40-50 for hypertrophic/keloid scars) and multiplied by the number of lesions, graded on a 4-point scale: 0 = none; 1 = <5 scars; 2 = 5-20 scars; 3 = >20 scars. The global score ranges from 0 to 540, with higher scores indicating greater severity. In this study, participants with hypertrophic or keloid scars will be excluded; therefore, only atrophic scar subtypes will be scored (subcategory 1).
ECCA grading scale (échelle d'évaluation clinique des cicatrices d'acné) | Assessments will be performed by blinded evaluators using standardized photographs at 16 weeks after the last session.
  The ECCA is a validated scale that quantifies acne scars through both qualitative and quantitative components. Scar type is weighted by a numerical factor (15-30 for atrophic scars and elastosis; 40-50 for hypertrophic/keloid scars) and multiplied by the number of lesions, graded on a 4-point scale: 0 = none; 1 = <5 scars; 2 = 5-20 scars; 3 = >20 scars. The global score ranges from 0 to 540, with higher scores indicating greater severity. In this study, participants with hypertrophic or keloid scars will be excluded; therefore, only atrophic scar subtypes will be scored (subcategory 1).

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | From baseline to 30 days after the end of the treatment
  Blinded evaluators will perform side-by-side comparisons of baseline vs. 30-day photographs. Improvement will be graded on a 5-point ordinal scale.
Global Aesthetic Improvement Scale (GAIS) | From baseline to 16 weeks after the end of the treatment
  Blinded evaluators will perform side-by-side comparisons of baseline vs. 16 weeks photographs. Improvement will be graded on a 5-point ordinal scale.
Goodman & Baron Acne Scar Scale | Baseline
  Scars will be categorized according to morphology, recording the number of mild, moderate, severe, and hypertrophic lesions. An algorithm will generate a total score (range: 0-84), with higher scores indicating greater severity and number of scars. This scoring system reflects both the type and frequency of lesions, with higher values representing worse scar severity.
Goodman & Baron Acne Scar Scale | 30 days after the end of the treatment
  Scars will be categorized according to morphology, recording the number of mild, moderate, severe, and hypertrophic lesions. An algorithm will generate a total score (range: 0-84), with higher scores indicating greater severity and number of scars. This scoring system reflects both the type and frequency of lesions, with higher values representing worse scar severity.
Goodman & Baron Acne Scar Scale | 16 weeks after the end of the treatment
  Scars will be categorized according to morphology, recording the number of mild, moderate, severe, and hypertrophic lesions. An algorithm will generate a total score (range: 0-84), with higher scores indicating greater severity and number of scars. This scoring system reflects both the type and frequency of lesions, with higher values representing worse scar severity.
Improvement perceived by patients | 30 days after the end of the treatment
  articipants will self-assess their improvement using a quartile grading scale. This measure captures the subjective satisfaction of the participant and complements the blinded clinical assessments.
Satisfaction reported by patient | 30 days after the end of the treatment
  Satisfaction reported by Likert scale.
Downtime | From the day after each treatment session until up to 9 days post-treatment.
  Recovery time will be recorded in days and defined as the period in which the participant experiences visible clinical signs (such as erythema or edema) and local discomfort (burning, pain, or itching), leading to physical or aesthetic limitations. Participants will complete a standardized daily questionnaire, administered via telephone contact by the study investigator, to report the presence of symptoms and whether they avoided public activities due to skin appearance. This outcome aims to quantify, in a subjective and functional way, the short-term impact of treatment on quality of life, social activities, and overall tolerability.
Pain - Visual Analog Scale (VAS) | Immediately after each treatment session.
  Pain will be assessed using the Visual Analog Scale (VAS), a 10-cm straight line where 0 represents "no pain" and 10 represents "worst possible pain." Immediately after each session, participants will be asked to mark the point on the line that best represents the pain experienced during the procedure.
Adverse Events | Daily for 10 days after each treatment session.
  Participants will be contacted daily via WhatsApp message or phone call to report the presence or absence of adverse events, including pain, erythema, edema, infection, discharge, crusts, hyperpigmentation, or scarring.
Adverse Events | Weekly until 30 days after the last treatment session.
  Participants will be contacted daily via WhatsApp message or phone call to report the presence or absence of adverse events, including pain, erythema, edema, infection, discharge, crusts, hyperpigmentation, or scarring.
Adverse Events | 60 days after the last treatment session.
  Participants will be contacted daily via WhatsApp message or phone call to report the presence or absence of adverse events, including pain, erythema, edema, infection, discharge, crusts, hyperpigmentation, or scarring.
Adverse Events | 90 days after the last treatment session.
  Participants will be contacted daily via WhatsApp message or phone call to report the presence or absence of adverse events, including pain, erythema, edema, infection, discharge, crusts, hyperpigmentation, or scarring.
Facial Acne Scar Quality of Life - FASQoL | Baseline
  A ten questions instrument, presenting 5 answers for each question, giving 0-4 points. A total of 0-40 points will be find, being higher the higest impact in quality of life.
Facial Acne Scar Quality of Life - FASQoL | 30 days after the end of the treatment
  A ten questions instrument, presenting 5 answers for each question, giving 0-4 points. A total of 0-40 points will be find, being higher the higest impact in quality of life.
Dermatology Life Quality index DLQI | Baseline
  The Dermatology Life Quality Index (DLQI) is a 10-question, self-administered questionnaire for adults (16+) to measure the impact of skin disease on their daily lives over the past week.
Dermatology Life Quality index DLQI | 30 days after the end of the treatment
  The Dermatology Life Quality Index (DLQI) is a 10-question, self-administered questionnaire for adults (16+) to measure the impact of skin disease on their daily lives over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Pavani, PhD, Study Chair — University of Nove de Julho; Luciana Khachikian, Master Student, Principal Investigator — University of Nove de Julho
Locations (1):
- Espaço Conceito Medical San, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All colected IPD will be shared, except individual photographs.
Supporting Information: SAP
Time Frame: The IPD will be available after the publication of the results, for 10 years.
Access Criteria: The IPD will be available as a excel file.